CLINICAL TRIAL: NCT02175524
Title: The Association Between Areca-nut Chewing Habit and Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CF13341
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Oral and Esophageal Cancer; Metabolic Syndrome.
Keywords: nut chewing
MeSH Terms: conditions — Esophageal Neoplasms; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Patients proved to be oral and esophageal cancer and had the habit of areca nut chewing.
- Control: Patients proved to be oral and esophageal cancer and did not have the habit of areca nut chewing.

SUMMARY:
The purpose of this study is going to determine the odds ratio of metabolic syndrome (MS), the habit of areca nut chewing, antioxidant, and inflammatory status in oral and esophageal patients. The current study was designed as a case-control study. Patients proved to be oral and esophageal cancer and had the habit of areca nut chewing are defined as case group. Patients proved to be oral and esophageal cancer and did not have the habit of areca nut chewing are defined as control group. The participants' age, blood pressures, and smoking habits will be recorded. Body weight, height, waist, and hip circumferences will be measured. Fasting venous blood samples will be obtained to determine hematological parameters [i.e., serum creatinine, total cholesterol, triacylglycerol, low density lipoprotein-cholesterol, high density lipoprotein-cholesterol, malondialdehyde, superoxide dismutase, glutathione peroxidase, catalase, and inflammatory markers (C-reactive protein, tumor necrosis factor-alpha, and interleukin-6)]. Logistic regression analyses are going to perform to examine the relationship between areca nut chewing and MS in this population. If we can make sure the relationship between areca nut chewing and MS, the clinicians and nutritionists can teach people to quit areca nut chewing in order to avoid the possibility of developing metabolic syndrome and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients proved to be oral and esophageal cancer will be recruited.

Exclusion Criteria:

* Subjects with diabetes mellitus, liver, renal diseases, or undergoing statin therapy.
* Taking antioxidant vitamins supplements.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with oral and oesophageal carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Metabolic syndrome | Up to 1 week
  Measure blood pressure, blood lipid profiles, fasting glucose, and waist circumferences.

SECONDARY OUTCOMES:
Antioxidant activity | Up to 1 week
  Antioxidant ability measurements: lipid peroxidation markers (MDA), antioxidant enzymes activities (catalase, glutathione peroxidase, and superoxide dismutase).
Inflammatory status | Up to 1 week
  Measure inflammatory markers: C-reactive protein, Interleukin-6, and tumor necrosis factor-alpha.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Verterans General Hospital, Taichung, Taiwan